CLINICAL TRIAL: NCT00324415
Title: Phase II Trial of Combined Modality Therapy Plus Cetuximab in HIV-Associated Anal Carcinoma
Brief Title: Combined Modality Therapy for Patients With With HIV and Stage I, Stage II, or Stage III Anal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-045; U01CA070019 (NIH); CDR0000440065 (Other: NCI)
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Results first posted 2015-09-17 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Anal Cancer
Keywords: stage I anal cancer; stage II anal cancer; stage IIIA anal cancer; stage IIIB anal cancer; squamous cell carcinoma of the anus; basaloid carcinoma of the anus; cloacogenic carcinoma of the anus
MeSH Terms: conditions — Anus Neoplasms; Anal Canal Carcinoma | interventions — Cetuximab; Cisplatin; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CMT with Radiation Therapy (Experimental): All patients will receive combined modality therapy (CMT) with 2 cycles of cisplatin and 5-FU chemotherapy, given concurrently with radiation therapy. CMT consists of:
  * Cetuximab 400 mg/m2 IV Day -7 (1 week before the cycle 1, Day 1 cisplatin/5-FU and RT), then 250 mg/m2 IV Days 1, 8, 15, 22, 29, 36 and 43 (a minimum of 6 and a maximum of 8 doses of cetuximab will be administered, including the loading dose).
  * Cisplatin 75 mg/m2 IV on Day 1 (cycle 1) and Day 29 (cycle 2)
  * 5-FU 1000 mg/m2/day by continuous intravenous infusion on Days 1-4 (cycle 1) and Days 29-32 (cycle 2)
  Interventions: Biological: cetuximab; Drug: cisplatin; Drug: fluorouracil; Radiation: radiation therapy

INTERVENTIONS:
Biological: cetuximab — 400 mg/m2 IV Day -7 (1 week before the cycle 1, Day 1 cisplatin/5-FU and RT), then 250 mg/m2 IV Days 1, 8, 15, 22, 29, 36 and 43 (a minimum of 6 and a maximum of 8 doses of cetuximab will be administered, including the loading dose)
  Other Names: Erbitux
Drug: cisplatin — 75 mg/m2 IV on Day 1 (cycle 1) and Day 29 (cycle 2)
  Other Names: Platinol
Drug: fluorouracil — 1000 mg/m2/day by continuous intravenous infusion on Days 1-4 (cycle 1) and Days 29-32 (cycle 2)
  Other Names: 5-FU; Adrucil; Carac; Efudex; Fluoroplex
Radiation: radiation therapy — Irradiation to tumor site and inguinal nodes beginning on cycle 1, Day 1 cisplatin/5-FU (minimum 45.0 Gy [5 weeks if given on schedule and without interruption], maximum 54.0 Gy [6 weeks if given on schedule and without interruption). IMRT may be used at the discretion of the treating physician.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving cisplatin, fluorouracil, and cetuximab together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cisplatin, fluorouracil, and cetuximab together with radiation therapy works in treating patients with HIV and stage I, stage II, or stage III anal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 2-year local failure rate in patients with HIV-associated stage I-IIIB anal carcinoma treated with cisplatin, fluorouracil, cetuximab, and radiotherapy.
* Determine the objective response rate (complete and partial), progression-free survival, relapse-free survival, colostomy-free survival, overall survival, quality of life, and overall toxicity in patients treated with this regimen.

Secondary

* Characterize the effect of this regimen on the underlying HIV condition by describing changes in viral load, CD4 counts, and the incidence of opportunistic illnesses, including the development of AIDS during and in the first year after treatment.
* Evaluate the effect of this regimen on anogenital human papilloma virus (HPV) infection and anal cytology.

OUTLINE: This is an open-label, multicenter study.

Patients receive cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, and 35*, fluorouracil IV continuously on days 1-4 and 29-32, and cisplatin IV over 1 hour on days 1 and 29. Beginning on day 1, patients undergo concurrent radiotherapy to the primary tumor 5 days a week for 5-7 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients receiving 7 weeks of radiotherapy also receive cetuximab on days 42 and 49.

Quality of life is assessed at baseline, at the completion of study treatment, and then at months 3, 6, 12, 24, and 36.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 47 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage I-IIIB invasive anal canal or perianal (anal margin) squamous cell carcinoma, including tumors with any of the following nonkeratinizing histologies:

  * Basaloid
  * Transitional cell
  * Cloacogenic
* Documented HIV infection by 1 of the following:

  * Antibody detection
  * Culture
  * Quantitative assay of plasma HIV RNA

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL (transfusions, epoetin alfa, or myeloid growth factor support allowed provided blood counts are stable for ≥ 2 weeks prior to study entry)
* Creatinine ≤ 1.5 times upper limit of normal (ULN) OR creatinine clearance > 60 mL/min
* AST and ALT ≤ 3 times ULN
* Bilirubin ≤ 2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No acute active, serious, uncontrolled opportunistic infection
* No other prior invasive malignancy diagnosed within the past 24 months, excluding in situ cervical cancer, anal dysplasia or carcinoma in situ, nonmelanoma skin carcinoma, or Kaposi's sarcoma that has not required systemic chemotherapy within the past 24 months
* No peripheral neuropathy > grade 1
* No severe or poorly controlled diarrhea
* No medical or psychiatric illness that would preclude study requirements

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for this malignancy

  * Prior radiotherapy for another condition (e.g., Kaposi's sarcoma) allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-09; Primary Completion 2014-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A. Sparano, MD, Study Chair — Albert Einstein College of Medicine; Lisa A. Kachnic, MD, Principal Investigator — Massachusetts General Hospital; David M. Aboulafia, MD, Principal Investigator — Floyd & Delores Jones Cancer Institute at Virginia Mason Medical Center
Locations (7):
- United States (7):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Benaroya Research Institute at Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Result] Sparano JA, Lee JY, Palefsky J, Henry DH, Wachsman W, Rajdev L, Aboulafia D, Ratner L, Fitzgerald TJ, Kachnic L, Mitsuyasu R. Cetuximab Plus Chemoradiotherapy for HIV-Associated Anal Carcinoma: A Phase II AIDS Malignancy Consortium Trial. J Clin Oncol. 2017 Mar;35(7):727-733. doi: 10.1200/JCO.2016.69.1642. Epub 2016 Dec 12. PMID 27937092

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Modality Therapy: Combined modality therapy consists of cisplatin, 5-flourouracil, and irradiation plus cetuximab
Period: Overall Study
Arm/Group | Combined Modality Therapy
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Combined Modality Therapy: cisplatin, 5-flourouruacil, and irradiation plus cetuximab.
Arm/Group | Combined Modality Therapy
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 28
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Locoregional Failure Rate at 3 Years
Description: Patients will be classified into two groups for purposes of primary endpoint analysis: failure or no failure at 3 years (in the primary analysis, patients lost to follow-up prior to 3 years will be considered failures). For the secondary endpoint of objective response, patients will be classified as responders
Time Frame: 3 years following completion of therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined Modality Therapy
Number analyzed (Participants) | 45
percentage of participants
  LRF rate by including censored patients treated as failures | 42 [28 to 56]
  LRF rate as per Kaplan-Meier estimate | 20 [10 to 37]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival at 1 year is the percentage of patients who are alive and have not experienced progressive disease, defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started, or the appearance of one or more new lesions.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined Modality Therapy
Number analyzed (Participants) | 45
percentage of participants | 87.3 [72.1 to 94.5]

3. Secondary Outcome: Relapse-free Survival
Description: Percentage of participants who are alive and have not experienced progressive disease and have not relapsed
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined Modality Therapy
Number analyzed (Participants) | 45
percentage of participants | 83.1 [67.8 to 91.6]

4. Secondary Outcome: Colostomy-free Survival at 1 Year
Description: Percentage of participants who are alive and have not had a colostomy
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined Modality Therapy
Number analyzed (Participants) | 45
percentage of participants | 92.4 [78.3 to 97.5]

5. Secondary Outcome: Overall Survival
Description: Percentage of participants who are alive at one year
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined Modality Therapy
Number analyzed (Participants) | 45
percentage of participants | 92.8 [79.4 to 97.7]

6. Secondary Outcome: Quality of Life EORTC Global Score at 1 Year
Description: EORTC QLQ-C30 Global Score at 1 year. The EORTC QLQ-C30 is a validated questionnaire that evaluates quality of life. The global score is an overall score for quality of life that ranges from 0 to 100. Higher scores indicate between quality of life
Time Frame: 1 year
Population: The number of participants analyzed is the number of participants for whom quality of life questionnaires were completed at one year.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Modality Therapy
Number analyzed (Participants) | 29
units on a scale | 78.9 (24.0)

7. Secondary Outcome: Number of Delayed Toxicities
Description: Delayed toxicities are defined as toxicities that occur over 90 days following treatment completion
Time Frame: 90 days following treatment discontinuation
Measure: Number; unit: events
Arm/Group | Combined Modality Therapy
Number analyzed (Participants) | 45
events | 5

8. Secondary Outcome: Changes in CD4 Counts During and for 1 Year After Completion of Study Treatment
Description: Change in absolute CD4 counts from start of treatment to 1 year after completion of study treatment
Time Frame: 1 year following treatment discontinuation
Population: The number of participants analyzed is the number for whom absolute CD4 count data were available at baseline at at 1 year after study completion
Measure: Median (Full Range); unit: cells/mm3
Arm/Group | Combined Modality Therapy
Number analyzed (Participants) | 38
cells/mm3 | 102 [-403 to 669]

9. Secondary Outcome: Incidence of Opportunistic Illnesses
Description: Incidence of opportunistic illnesses, including the development of AIDS during and for 1 year after completion of study treatment
Time Frame: 1 year following treatment discontinuation
Measure: Number; unit: participants
Arm/Group | Combined Modality Therapy
Number analyzed (Participants) | 45
participants | 4

10. Secondary Outcome: Objective Response Rate (Complete and Partial)
Description: Number of participants with complete and partial responses based on the RECIST criteria
Time Frame: 3 years following treatment discontinuation
Measure: Number; unit: participants
Arm/Group | Combined Modality Therapy
Number analyzed (Participants) | 45
participants | 30

11. Other Pre Specified Outcome: Count of Participants by Type of HPV at Baseline
Description: Descriptive statistics will be used to describe the types of HPV found in baseline anal swabs and tissue biopsies.
  Proportion of cases with each type will be summarized
Time Frame: baseline
Population: Participants with available HPV status data
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Modality Therapy
Number analyzed (Participants) | 30
Participants
  HPV 16 | 16
  HPV 6 | 9
  HPV 11 | 9
  HPV 18 | 5
  HPV 31 | 5
  HPV 33 | 3
  HPV 82 | 3
  HPV 68 | 3
  HPV 51 | 2
  HPV 52 | 2
  HPV 26 | 1
  HPV 30 | 1
  HPV 32 | 1
  HPV 35 | 1
  HPV 45 | 1
  HPV 54 | 1
  HPV 53 | 1
  HPV 56 | 1
  HPV 58 | 1
  HPV 69 | 1
  HPV 72 | 1
  HPV 73 | 1
  HPV 86 | 1
  HPV 87 | 1
  HPV 97 | 1
  Mixed | 1

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Combined Modality Therapy
Serious Adverse Events (participants affected / at risk) | 27/45
Other Adverse Events (participants affected / at risk) | 41/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Modality Therapy (N=45)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Anal fistula (Gastrointestinal disorders) | 2 (2)
Anal mucositis (Gastrointestinal disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 8 (9)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Oral mucositis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
death NOS (General disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Anorectal infection (Infections and infestations) | 3 (3)
Lung infection (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Scrotal infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Radiation reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 3 (3)
White blood count decreased (Investigations) | 3 (3)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 9 (9)
Hypokalemia (Metabolism and nutrition disorders) | 9 (9)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Metabolism and nutrition disorders) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
melena (Gastrointestinal disorders) | 1 (1)
Infection with grade 3 or 4 neutrophils (Infections and infestations) | 2 (2)
Lung pneumonia (Infections and infestations) | 1 (1)
Toxoplasmosis with Hydrocephalus (Infections and infestations) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other skin disorder (Skin and subcutaneous tissue disorders) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Modality Therapy (N=45)
Anemia (Blood and lymphatic system disorders) | 14 (26)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 7 (7)
Anal pain (Gastrointestinal disorders) | 10 (14)
Diarrhea (Gastrointestinal disorders) | 22 (38)
Other GI disorders (Gastrointestinal disorders) | 9 (21)
Oral mucositis (Gastrointestinal disorders) | 10 (23)
Nausea (Gastrointestinal disorders) | 12 (18)
Proctitis (Gastrointestinal disorders) | 5 (7)
Rectal pain (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 7 (8)
Fatigue (General disorders) | 17 (18)
Fever (General disorders) | 5 (5)
Other blood and lymphatic disorders (Blood and lymphatic system disorders) | 5 (7)
Other general disorders (General disorders) | 6 (7)
Pain (General disorders) | 3 (4)
Anorectal infection (Infections and infestations) | 3 (3)
Other infections (Infections and infestations) | 4 (6)
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 (3)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 11 (16)
Alanine aminotransferase increased (Investigations) | 4 (4)
Aspartate aminotransferase increased (Injury, poisoning and procedural complications) | 4 (4)
Blood bilirubin increased (Investigations) | 3 (6)
Neutrophil count decreased (Investigations) | 10 (18)
Platelet count decreased (Investigations) | 13 (17)
Weight loss (Investigations) | 11 (12)
White blood cell decreased (Investigations) | 11 (34)
Anorexia (Metabolism and nutrition disorders) | 9 (11)
Dehydration (Metabolism and nutrition disorders) | 10 (11)
hypoalbuminemia (Metabolism and nutrition disorders) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (9)
Hypokalemia (Metabolism and nutrition disorders) | 10 (17)
Hypomagnesia (Metabolism and nutrition disorders) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 7 (11)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Anxiety (Nervous system disorders) | 3 (3)
Depression (Nervous system disorders) | 4 (4)
Insomnia (Nervous system disorders) | 4 (4)
Other renal and urinary disorders (Renal and urinary disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 12 (15)
Other skin disorders (Skin and subcutaneous tissue disorders) | 12 (20)
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT00324415/Prot_SAP_001.pdf